CLINICAL TRIAL: NCT07206901
Title: Evaluation of an Ayurvedic Herbal Compound (Maharishi Amrit Kalash) Compared to Vitamins C+E and Placebo on Vascular Function in High CVD Risk Subjects: A Randomized Controlled Trial
Brief Title: Evaluation of an Ayurvedic Herbal Compound Compared to Vitamins C+E and Placebo on Vascular Function in High-Risk Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi International University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Howard University (Other)
Responsible Party: Principal Investigator, Robert Schneider, MD, Director and Professor, Maharishi International University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HH2100mdjs; P50AT000082 (NIH)
Record Dates: First submitted 2025-09-05; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease
Keywords: brachial artery reactivity (BART); Maharishi Amrit Kalash (MAK); herbal preparation; Ayurvedic herbal preparation; vascular function
MeSH Terms: conditions — Coronary Artery Disease | interventions — Maharishi Amrit Kalash; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: randomized double blind placebo controlled trial with two active groups and a placebo control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ayurvedic herbal compound (Experimental): Maharishi Amrit Kalash (MAK) is an Ayurvedic herbal compound classified as a Rasayana. MAK is a commercially available product that can be purchased and consumed in paste or tablet form. For this double blind study, MAK was administered in tablet form.
  Interventions: Dietary Supplement: Maharishi Amrit Kalash
- vitamin supplement (Active Comparator): Vitamin C and E combination supplement. For this study, it was manufactured with the same shape and color as experimental tablet (MAK)
  Interventions: Dietary Supplement: vitamin C + E
- placebo (Placebo Comparator)
  Interventions: Other: Inert Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Maharishi Amrit Kalash
  Arms: Ayurvedic herbal compound
Dietary Supplement: vitamin C + E
  Arms: vitamin supplement
Other: Inert Placebo Capsule — placebo is same shape and color as is the active interventions but is inert
  Arms: placebo

SUMMARY:
This was a randomized controlled trial aimed to evaluate the effects of an herbal Ayurvedic herbal supplement in comparison to a Vitamin C/E supplement and an inert placebo on heart health. There were three treatment groups: Maharishi Amrit Kalash (MAK), vitamin C+E and the placebo group. The primary outcome was smooth muscle responsiveness, blood flow and dilation using the brachial artery reactivity test in a Black population at risk for heart disease.

DETAILED DESCRIPTION:
This was a randomized placebo controlled clinical trial that recruited 143 urban Black men and women at risk for cardiovascular disease (CVD) in the Washington, DC and surrounding areas. Participants were randomly assigned to one of three treatment groups: Maharishi Amrit Kalash (MAK), Vitamin C and E supplement (VitCE) or placebo. The intervention period was 12 months.

Study inclusion criteria was the following: Black (self-identified), atherosclerotic coronary heart disease defined by a clinical history of myocardial infarction, coronary revascularization procedure (CABG or coronary angiography with at least one artery showing >50% stenosis, or > 2 points on the ATP III risk factor scale, informed consent and permission from patients physician. Exclusion criteria included decompensated heart failure, renal or hepatic insufficiency, or contraindications to nitroglycerin. Participants provided written informed con-sent. Institutional review board approval was obtained.

All nutritional supplements (i.e. treatments) used in this study were available in white plastic bottles, sealed and capped. Each Participant received one pair of bottles (one yellow and one green) at each clinic visit every two months. All pills were coated white and were manufactured in tablet form to more easily conceal the participants treatment status.

Clinical measures included brachial artery reactivity (BART) testing, carotid intima medial thickness (cIMT) assessment and blood pressure and lipid level monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Ethnicity: African American, self-identified
* Age: 55 years and older
* Medically documented coronary artery disease (CAD/CHD): defined by previous myocardial infarction OR revascularization procedure-coronary artery bypass grafting (CABG), or percutaneous transluminal coronary angioplasty (PCTA), OR coronary angiography with at least one coronary artery with > 50% stenosis.
* In the absence of documented CAD/CHD above, then at least two risk factor points on the Framingham/ATPIII risk factor scoring assessment.
* Signed informed consent
* Permission of Participant's primary physician (if feasible)

Exclusion Criteria:

* Myocardial infarction, unstable angina, coronary artery by-pass grafting (CABG), percutaneous transluminal coronary angioplasty (PTCA), or stroke within preceding three months.
* Carotid artery endarterectomy.
* Arrhythmia atrial fibrillation, second or third degree AV block.
* Congestive heart failure-Class III or IV or ejection fraction less than 30 percent.
* Clinically significant valvular heart disease.
* Clinically significant hepatic or renal failure.
* Major psychiatric disorders, current alcohol/dependency disorder, or other drug abuse dependency disorder.
* Non-cardiac life threatening illness.
* Participating in a formal stress management program.
* Plans to move out of the study area or travel extensively.
* Unwillingness to accept randomization into any study group.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2002-10-14 (Actual); Primary Completion 2006-07-31 (Actual); Study Completion 2014-10-27 (Actual)

PRIMARY OUTCOMES:
Brachial Artery Reactivity | 0 months and 12 months
  This is a clinical test or protocol that measures the reactivity of the brachial artery and its ability to vasodilate in response to increased blood flow, typically assessed using ultrasound imaging. It is administered with a hyperemia phase (occlusion of the right arm with a cuff) followed by release and/or a sublingual nitroglycerin phase in which a small dose of nitroglycerin is placed under the tongue of the patient in a supine position. In each case, the flow mediated dilation (FMD) of the brachial artery is measured as a marker of vascular health.

SECONDARY OUTCOMES:
carotid intima medial thickness | 0 and 12 months
  B mode doppler ultrasound measurement of the carotid artery
blood pressure | 0 and 12 months
  clinical assessment of systolic and diastolic blood pressure
lipid profile | 0 and 12 months
  laboratory assessment of blood levels of cholesterol, LDL, HDL and triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Schneider, MD, Principal Investigator — Maharishi International University
Locations (1):
- College of Integrative Medicine, Fairfield, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
raw data can be shared along with Participant ID codes but not full names, initials or contact information about the study participants